CLINICAL TRIAL: NCT01369966
Title: Brain Circuits in Schizophrenia and Smoking
Status: Completed | Type: Observational
Sponsor: National Institute on Drug Abuse (NIDA) (NIH)
Responsible Party: Sponsor
Organization: National Institutes of Health Clinical Center (CC) (NIH)
Other Study IDs: 999911467; 11-DA-N467
Record Dates: First submitted 2011-06-08; First posted 2011-06-09 (Estimated); Last update posted 2018-04-05 (Actual); Status verified 2014-12-24

CONDITIONS: Schizophrenia; Smoking Cessation; Nicotine Abuse
Keywords: Smoking Cessation; Schizophrenic Smokers; fMRI; Neural Circuits
MeSH Terms: conditions — Schizophrenia; Smoking Cessation

STUDY DESIGN:
Time Perspective: Other

SUMMARY:
Background:

- Smoking is associated with serious health risks. People who have mental illness are more likely to smoke. Researchers are studying the brain circuits linked with smoking and nicotine craving. This study will look at whether a specific brain circuit can explain the high rate of smoking in people with schizophrenia.

Objectives:

- To study brain activity in smokers and nonsmokers with and without schizophrenia, as well as their family members.

Eligibility:

* Current smokers (at least 100 cigarettes in the past year) and nonsmokers between 18 and 62 years of age in one of the following groups:
* Have been diagnosed with schizophrenia.
* Family members of those with schizophrenia.
* Healthy adults with no history of severe mental illness or brain trauma.
* Family members of the healthy adults.

Design:

* People in the study will be screened with a physical exam, medical history, questionnaires, and blood tests.
* They will have up to three visits: the screening visit and two study visits (each given 1 year apart).
* At the first study visit, those taking part will be trained in the tests they will do during the magnetic resonance imaging (MRI) scan. Then they will have the MRI scan.
* After the first study visit, current smokers will receive phone calls from the study researchers every other month for 1 year. They will be asked about their smoking habits.
* At the second study visit, current smokers and some nonsmokers will have another MRI scan and the same tests as before.
* Current smokers will receive a final phone call 1 year after the second study visit. They will be asked to give information about their smoking habits.

DETAILED DESCRIPTION:
Objective

The health risk associated with tobacco use is high, and is even higher in people with severe mental illness. The underlying brain circuitry for smoking-mental illness comorbidity is unknown. Identifying brain comorbidity circuitry is important for new therapeutic development. This study will examine whether a specific brain circuitry can explain the high rate of smoking in patients with schizophrenia. Identifying the key brain circuits associated with smoking, especially smoking in a high risk population, will provide concrete biomarkers for new therapeutic development, and ultimately reducing the smoking related health burden.

Study Population

Schizophrenic patients and their family members, non-schizophrenia controls and their family members, including smokers and nonsmokers in each of the four groups will be included in this study.

Design

1. A cross-sectional study for all subjects at baseline. They will receive clinical and diagnostic interviews, functional, symptom, and cognitive testing, and MRI. They will also have blood drawn, to identify brain circuits and covariates associated with the severe smoking problem in schizophrenia.
2. A prospective longitudinal study design where smokers will be encouraged to quit smoking and smoking cessation support is provided if needed, followed by retesting of imaging and some clinical assessments, to identify brain circuits associated smoking cessation or the difficulty of quitting in schizophrenia and non-schizophrenia smokers.

Outcome Measures

Combining event-related and resting fMRI techniques, we propose to test the hypothesis that an abnormal dorsal anterior cingulate cortex (dACC) and ventral striatum (VS) circuit underlies the high prevalence of comorbid smoking in schizophrenia. We also propose to test specific clinical implications of this circuit including a within-subject event-related fMRI study to test the mechanistic implication of the rsFC signals, a prospective follow-up to test the circuit s predictive validity on smoking behavior change, and genetic studies to describe the path from genes to brain circuits to smoking behaviors.

ELIGIBILITY:
* INCLUSION CRITERIA:

For all participants (patients, healthy controls, and family members):

1. Male and Female between ages 18-62
2. Ability to give written informed consent

For patients (smokers and non-smokers)

1. Must have a DSM-IV diagnosis of schizophrenia, schizoaffective disorder, or schizophreniform disorder.
2. Must be clinically stable in the opinion of the patient s treating clinician with no change in antipsychotic medications or any dosage adjustment for 2 weeks or more preceding study enrollment as well as 2 weeks or more prior to each of the MRI scans.

For smokers (patients, healthy controls, and family members):

1. Must have smoked at least 100 cigarettes in the last year and currently smoking daily (at any amount).

For family members only:

1. Have a least one first-degree family member who is eligible for participating in this protocol as a patient or a smoker as defined above

EXCLUSION CRITERIA:

For patients only:

1. Evaluation to Sign Consent (ESC) score below 12.

For all participants (patients and healthy controls):

1. Any medical illnesses that may affect normal brain functioning, based on the screening history. Examples of these conditions include, but not limited to, stroke, repeated seizure, history of significant head trauma, CNS infection or tumor, other significant brain neurological conditions.
2. Substance dependence within 6 months or substance abuse within 1 month, other than nicotine or marijuana dependence.
3. Pregnancy
4. Cannot refrain from using alcohol and marijuana for 24 hours
5. Unable to safely undergo MRI scanning due to metallic devices or objects (cardiac pacemaker or neurostimulator, some artificial joints, metal pins, surgical clips or other implanted or non-removable metal parts), claustrophobic to the scanner, or unable to lie comfortably supine for up to 2 hours
6. Cannot safely give 70 ml blood based on the screening evaluation

For family members:

Family members meeting exclusion criteria 1-5 above may participate in the study unless they cannot safely give 70 ml blood. Their participation will, however, be limited to research interviews and questionnaires and phlebotomy or saliva collection for genetic testing.

Ages: 18 Years to 62 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 42 (Actual)
Dates: Start 2011-05-16; Study Completion 2014-12-24

PRIMARY OUTCOMES:
Test the hypothesis that dorsal anterior cingulate cortex - ventral straitum (dACC-VS) resting state functional connectivity (rsFC) is related to smoking in NC smokers and NC nonsmokers.

SECONDARY OUTCOMES:
Test the hypothesis that dACC-VS rsFC is associated with SZ by comparing SZ smokers and SZ nonsmokers with NCs above. First-degree relatives of SZ smokers will be included to rule out medication effects.
Examine the mechanistic implication of the rsFC measure using parallel resting & behavioral/cognitive task based fMRI; compare fMRI signals and test the hypothesis that reward/inhibition nodes/circuits and rsFC are associated with aspect...

CONTACTS AND LOCATIONS:
Overall Officials: Elliot Stein, Ph.D., Principal Investigator — National Institute on Drug Abuse (NIDA)
Locations (1):
- Maryland Psychiatric Research Center (MPRC) 55 Wade Avenue, Catonsville, Maryland, United States

REFERENCES:
- [Background] Abi-Dargham A, Gil R, Krystal J, Baldwin RM, Seibyl JP, Bowers M, van Dyck CH, Charney DS, Innis RB, Laruelle M. Increased striatal dopamine transmission in schizophrenia: confirmation in a second cohort. Am J Psychiatry. 1998 Jun;155(6):761-7. doi: 10.1176/ajp.155.6.761. PMID 9619147
- [Background] Aguilar MC, Gurpegui M, Diaz FJ, de Leon J. Nicotine dependence and symptoms in schizophrenia: naturalistic study of complex interactions. Br J Psychiatry. 2005 Mar;186:215-21. doi: 10.1192/bjp.186.3.215. PMID 15738502
- [Background] al'Absi M, Hatsukami D, Davis GL. Attenuated adrenocorticotropic responses to psychological stress are associated with early smoking relapse. Psychopharmacology (Berl). 2005 Aug;181(1):107-17. doi: 10.1007/s00213-005-2225-3. Epub 2005 Apr 15. PMID 15834539